CLINICAL TRIAL: NCT05781516
Title: A Prospective, Randomized Controlled Study to Compare the Efficacy and Safety of Baricitinib Combined With Glucocorticoid and Glucocorticoid Monotherapy in Proliferative IgG4-RD Patients With Eosinophilia
Brief Title: Baricitinib Plus Glucocorticoid for Eosinophilia in IgG4-RD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wen Zhang (Other)
Collaborators: Tongji Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor-Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Baricitinib for Eosinophilia
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: IgG4-related Disease With Eosinophilia
Keywords: IgG4-related disease; eosinophilia
MeSH Terms: conditions — Immunoglobulin G4-Related Disease; Eosinophilia | interventions — Prednisolone; baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone monotherapy (Placebo Comparator): Oral prednisolone 0.6-0.8mg/kg daily for 4 weeks, then tapered and withdrawal in 4 months.
  Interventions: Drug: Prednisolone
- Prednisolone plus Baricitinib (Experimental): Oral prednisolone 0.6-0.8mg/kg daily for 4 weeks, then tapered and withdrawal in 4 months. Oral Baricitinib 2mg daily for 12 months.
  Interventions: Drug: Prednisolone; Drug: Baricitinib

INTERVENTIONS:
Drug: Prednisolone — Oral prednisolone 0.6-0.8mg/kg daily for 4 weeks, then tapered and withdrawal in 4 months.
Drug: Baricitinib — Oral Baricitinib 2mg daily for 12 months.
  Arms: Prednisolone plus Baricitinib

SUMMARY:
Evaluation of efficacy and safety of Baricitinib combined with glucocorticoid in patients of IgG4-related disease with eosinophilia.

DETAILED DESCRIPTION:
This is a multicenter, 52-week prospective, randomized controlled study to compare the efficacy and safety of Baricitinib combined with glucocorticoid and glucocorticoid monotherapy in proliferative IgG4-RD patients with eosinophilia.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must meet the following diagnostic criteria of IgG4RD (2020): 1) and radiological features: One or more organs show diffuse or localized swelling or a mass or nodule characteristic of IgG4-RD. In single organ involvement, lymph node swelling is omitted. 2) serological diagnosis: Serum IgG4 levels greater than 135 mg/dl. 3) diagnosis diagnosis: Positivity for two of the following three criteria: a. Dense lymphocyte and plasma cell infiltration with fibrosis. b. Ratio of IgG4-positive plasma cells /IgG-positive cells greater than 40% and the number of IgG4-positive plasma cells greater than 10 per high powered field. c. Typical tissue fibrosis, particularly storiform fibrosis, or obliterative phlebitis.

   Patients fulfill (1) + (2) + (3) are diagnosed as definite IgD4RD; (1) + (2): possible IgG4RD; (1) + (3): probable IgG4RD. exclusion of other diseases.
2. Active IgG4-RD (Responder Index ≥ 2 points for each involved organ)
3. The counts of peripheral blood eosinophil cells ≥0.75×109/L

Exclusion Criteria:

1. Patients who is not able to discontinue GC
2. Pregnancy or breastfeeding or planning to get pregnant within 2 years
3. Received glucocorticoids, immunosuppressants, biological agents or JAK inhibitors within 3 months
4. Allergic to Baricitinib
5. Concomitant other autoimmune diseases
6. Malignancy
7. Chronic HBV infection, latent tuberculosis, or active infection
8. Server liver or renal dysfunction, or heart failure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The difference of recurrent rate of IgG4-RD between the two groups | 52 weeks
  Clinical recurrence definition: any item of IgG4-RD Responder Index ≥2 (without treatment), or ≥ 3 (with treatment) or new organ involvement; with or without elevated serum IgG4 levels.

SECONDARY OUTCOMES:
The time of recurrence | 0-52 weeks
  Clinical recurrence definition: any item of IgG4-RD Responder Index ≥2 (without treatment), or ≥ 3 (with treatment) or new organ involvement; with or without elevated serum IgG4 levels.
The changes of IgG4-related disease Responder Index | 52 weeks
  According to international multispecialty validation study of IgG4-related disease Responder Index (Version: 13, December, 2015), Responder Index ≥ 0, and higher scores mean a worse outcome.
The changes of blood Eosinophil cells | 52 weeks
  Percentages (%) and counts (109) of peripheral eosinophil cells
The changes of serum IgG levels | 52 weeks
  Level of serum IgG(g/L)
The changes of serum IgG4 levels | 52 weeks
  Level of serum IgG4(mg/dL)
The changes of serum hsCRP level | 52 weeks
  Level of serum high-sensitivity C-reactive protein level(mg/L)
The changes of ESR | 52 weeks
  Serum erythrocyte sedimentation rate(mm/h)
The percentages of adverse events | 52 weeks
  Adverse effect of drugs
The changes of PGA | 52 weeks
  Changes of patient global assessment from baseline, score (0-10, higher is worse)
The results of High-throughput analysis | 52 weeks
  The changes of results from baseline in High-throughput analysis, including GWAS, single cell sequencing of B cell receptor.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Bejing, China